CLINICAL TRIAL: NCT00360841
Title: Stimulation of Auricular Acupuncture-Point for Chemotherapy-Induced Nausea/Vomiting: A Prospective Randomized Double-blind Cross-over Study
Brief Title: Stimulation of Auricular Acupuncture-Point for Chemotherapy-Induced Nausea/Vomiting
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 9561702041
Record Dates: First submitted 2006-08-04; First posted 2006-08-07 (Estimated); Last update posted 2012-12-06 (Estimated); Status verified 2012-11

CONDITIONS: Cancer
Keywords: auricular; acupuncture
MeSH Terms: conditions — Neoplasms | interventions — Acupuncture, Ear

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- A (Experimental): The subjects in arms A and B will receive auricular acupuncture. The subjects in arms A will receive auricular acupuncture (at 2nd and 4th chemotherapy courses) as well as the sham auricular acupuncture (at the 3rd chemotherapy course).
  Interventions: Procedure: Auricular acupuncture; Procedure: Sham auricular acupuncture
- B (Sham Comparator): The subjects in arms A and B will receive auricular acupuncture. The subjects in arm B will receive the sham auricular acupuncture (at the 2nd and 4th chemotherapy courses) and auricular acupuncture (at the 3rd chemotherapy course).
  Interventions: Procedure: Auricular acupuncture; Procedure: Sham auricular acupuncture
- C (No Intervention): No treatment received.

INTERVENTIONS:
Procedure: Auricular acupuncture — Subjects will be randomized to one of these arms. The subjects in arm A and B will receive auricular acupuncture. Before subjects receive chemotherapy within one day, they will be treated by auricular acupuncture, sham acupuncture, or control group.
  Arms: A; B
Procedure: Sham auricular acupuncture
  Arms: A; B

SUMMARY:
The purpose of this study is to evaluate auricular acupuncture as an antiemetic treatment compared with sham acupuncture and with no acupuncture in patients receiving moderately-high to highly emetogenic chemotherapy. Acupuncture constitutes a nonpharmacological intervention for chemotherapy-induced nausea/vomiting (CINV). Chinese medicine holds that stimulating select points both on the body and the ear, that lie along meridians or life channels, can relieve diseases.

DETAILED DESCRIPTION:
Chemotherapy-induced nausea and vomiting (CINV) are two of the most commonly reported adverse effects of chemotherapy. Uncontrolled CINV reduces quality of life, leads to delays in treatment, and causes serious metabolic disturbances. Current strategies for preventing acute CINV include combination therapy with a 5-HT3 antagonist and a corticosteroid for moderately-high to highly emetogenic chemotherapy. Similarly, strategies aimed at reducing the incidence and severity of delayed CINV include the combination of a corticosteroid and either a dopamine receptor antagonist or a 5-HT3 antagonist for 3-5 days post chemotherapy. Complete protection from vomiting in the first 24 hours is achieved in as many as 70-90% of patients receiving moderately-high and highly emetogenic chemotherapy; however, standard antiemetics only protect 50% of patients from experiencing nausea during this acute CINV phase. Delayed nausea and vomiting is less well defined and controlled, with as many as 50% of patients experiencing nausea and vomiting in the 3 to 5 day period following the first day of chemotherapy. Both acute and delayed CINV remain a significant problem in patients undergoing high-dose chemotherapy for autologous or allogeneic transplantation where up to 90% of patients experience CINV despite prophylactic strategies. Additional pharmacological interventions are clearly needed to optimize control of CINV. Neurokinin-1 receptor (NK-1) antagonists have been reported to improve the total control rates of acute CINV by approximately 25% compared to the standard combination of a 5-HT3 antagonists and dexamethasone alone. Cocquyt et al., reported that one dose of a NK-1 antagonist administered prior to cisplatin-based chemotherapy prevented delayed emesis in up to 72% of patients. Although promising, the role of these agents in CINV prevention and control is as yet undetermined. Acupuncture constitutes a nonpharmacological intervention for CINV. Chinese medicine holds that stimulating select points both on the body and the ear, that lie along meridians or life channels, can relieve diseases. From the previous studies, the P6 point, also known as the Neiguan point or G-Jo point no. 10, is located 2 cun (Chinese inch, equivalent to the width of an individual's thumb) proximal to the distal wrist crease, between the tendons of the palmaris longus and flexor carpi radialis. P6 acupuncture was shown to reduce the incidence and severity of nausea and vomiting in the postoperative setting, morning sickness, and the P6 transcutaneous electrical stimulation (TCES) therapy was shown to enhance the antiemetic action of ondansetron in patients receiving highly emetic chemotherapy treatment. Auricular acupuncture consisted of needle insertion in one ear at four points: (1) sympathetic - located in the terminal of the inferior antihelix crus; (2) stomach -located around the area where the helix crus terminates; (3) shinmoon - located at the bifurcating point between superior and inferior antihelix crus and the lateral 1/3 of the triangular fossa; and (4) occiput - located at the posterior superior corner of the lateral aspect of the antitragus have been reported to be effective in reducing PONV. The purpose of this study was to evaluate auricular acupuncture as an antiemetic treatment compared with sham acupuncture and with no acupuncture in patients receiving moderately-high to highly emetogenic chemotherapy.

The study is a three group, randomized, examiner-blind, crossover controlled trial. It is to evaluate the efficacy and safety of auricular acupuncture in patients receiving moderately-high to highly emetogenic chemotherapy from National Taiwan University Hospital. 120 eligible patients receiving moderately-high to highly emetogenic chemotherapy who fulfill the inclusion/exclusion criteria and complete the informed consent form will be recruited.

After the washout period of 2 weeks, the subjects will be required to take the medication for preventing acute CINV including combination therapy with a 5-HT3 antagonist and a corticosteroid for moderately-high to highly emetogenic chemotherapy. The patients will be divided into three groups (auricular acupuncture treatment group, sham auricular acupuncture treatment group, and non-treatment group) in order to test the effectiveness of auricular acupuncture. Group 1 patients will receive no treatment (control), after completion of the 1st chemotherapy course, Group 2 patients will receive auricular acupuncture treatment at the 2nd and 4th chemotherapy courses and will receive sham auricular acupuncture at the 3rd chemotherapy course, while Group 3 will receive sham auricular acupuncture at the 2nd and 4th chemotherapy courses and will receive auricular acupuncture at the 3rd chemotherapy course. At baseline visit and course 1, 2, 3, and 4 after chemotherapy, every subject will have efficacy evaluations by FILE, vomiting visual analog scare, WHOQOL-BREF questionnaire and Chinese Disposition Classification. Simultaneously, they will be monitored on their vital signs, complete blood counts, urinalysis, and biochemical indicators at baseline visit and the end of the trial. The collected data will then be analyzed by SAS 8.2 package.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed carcinoma
* Patients must have normal organ and marrow function as defined below:

  * ANC greater than or equal to 1500/mcL
  * Platelets greater than or equal to 100,000/mcL
  * AST (SGOT)/ALT (SGPT) less than 5 x institutional upper limit of normal
  * Creatinine within normal institutional limits, OR
  * Creatinine clearance greater than or equal to 60 mL/min/1.73 m2 for patients with creatinine levels less than 1.5mg/dl
* Patients should have the ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Patients with known CAD, CVA, epilepsy, hypotension, hypertension

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 103 (Actual)
Dates: Start 2006-06; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
At baseline visit and course 1, 2, 3, and 4 after chemotherapy, every subject will have been efficacy evaluated by FILE, vomiting visual analog scale, WHOQOL-Brief questionnaire and Chinese Disposition Classification. | subject

CONTACTS AND LOCATIONS:
Overall Officials: Chih-Hsin Yang, PhD, Principal Investigator — Deparment of Oncology, National Taiwan University Hospital
Locations (1):
- Department of Oncology, National Taiwan University Hospital, Taipei, Taiwan